CLINICAL TRIAL: NCT00590668
Title: Pulmonary Vein Ablation for Atrial Fibrillation: Safety Monitoring by Transesphoageal Echo, Intracardiac Echo and Computed Tomography and Assessment of Predictors of Recurrence and of Hypercoagulable State
Brief Title: Safety Monitoring of Patients Having Pulmonary Vein Ablation
Acronym: ROTEA
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Allan L. Klein, Principal Investigator, The Cleveland Clinic
Other Study IDs: 6104
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulmonary vein ablation; pulmonary vein stenosis
MeSH Terms: conditions — Atrial Fibrillation; Stenosis, Pulmonary Vein | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transesophageal Echocardiography — Measurement of peak diastolic flow velocity
  Other Names: TEE

SUMMARY:
Subjects eligible for this study have an irregular heartbeat called atrial fibrillation (AF)and who are scheduled for a procedure that involves applying electrical energy in your pulmonary veins, which is usually the site where this abnormal rhythm begins, or pulmonary vein ablation

We will examine the size and function of the left atrium (one of the 4 chambers of your heart) and the pulmonary veins before and after your ablation. This will be done by getting extra measurements during tests you will be having done which are ICE (intra cardiac echocardiography), TEE (transesophageal echocardiography) and CT scan (computed tomography), and drawing some blood samples.

The purpose of getting these extra measurements and blood samples is:

1. to see whether TEE measurements done before your ablation can tell us if your atrial fibrillation may come back after you ablation;
2. to see if TEE measurements look different before and after your ablation;
3. to see if a blood test can tell us if your atrial fibrillation may come back after your ablation;
4. to look at how often pulmonary vein narrowing is found by TEE compared to how often it is found by CT scan.

During the clinically indicated tests the doctor has ordered (TEE, ICE, CT scan), there will be additional measurements taken as a part of this research. This means that the TEE exam will last an additional 10-15 minutes, and the ICE procedure will last an additional 5-10 minutes. There is no additional time needed for the CT scan. In addition, we will be drawing 20 cc of blood (approximately four teaspoons).

The regularly scheduled follow up visit is usually three months after your ablation, we will again be getting some extra measurements from the TEE and CT scan. This will add about 10-15 minutes to the TEE test, but no additional time will be needed for the CT scan. In addition, we will be drawing 10 cc of blood drawn (approximately two teaspoons). A ventilation-perfusion scan of the lungs will also be performed as part of standard clinical care if significant PV stenosis is found by CT and/or TEE.

DETAILED DESCRIPTION:
Aims

1. Examine the structure and function of the left atrium, left atrial appendage and pulmonary veins before and after ablation.
2. Compare the findings of transesophageal echo with those from intracardiac echo.
3. Detect the incidence of pulmonary vein stenosis assessed by transesophageal echo compared to computed tomography.
4. Assess for physiological predictors for recurrence of atrial fibrillation based on echocardiography.
5. Determine whether biological markers such as B-type natriuretic peptide or C-reactive protein predict recurrence of atrial fibrillation.
6. Assess if markers of coagulation such as D-dimer and prothrombin factor 1.2 are increased in atrial fibrillation and could predict thromboembolic risk.

General Procedures Prior to ablation, blood will be drawn for measuring c-reactive protein, brain natriuretic polypeptide, D-dimer and prothrombin fragment 1.2. A transesopahegeal echocardiogram and an intracardiac echocardiogram will be performed. Then following sterile techniques, standard catheters will be passed through veins and positioned into the heart using X-ray guidance, and will cross the wall that divides the upper chambers of the heart so that the left atrium can be reached.The catheters will be used to trigger sites that originate the anomalous rhythm and once these are identified the generator will deliver radiofrequency energy to destroy the areas that cause irregular beats. After ablation follow-up visits will be done at one, three, six and twelve months. During that time several tests such as electrocardiograms, 24 hour Holter recording, computed tomography of the heart, transesophageal echocardiogram and repeated blood drawing to measure c-reactive protein, brain natriuretic peptide, D-dimer and prothrombin fragment 1.2 will be done.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or paroxysmal AF, resistanct to medical therapy
* Normal renal function (creatininine <1.5

Exclusion Criteria:

* Unable or unwilling to give informed consent
* History of esophageal diseases, such as stricture, vaices or cancer
* Inability to swallow TEE probe
* Severe mitral stenosis
* Severe mitral reguritation
* Cardiothoracic surgery within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonry vein ablation subjects at the Cleveland Clinic
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2004-05 (Actual); Primary Completion 2008-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
incidence of pulmonry vein stenosis following PVI | 3 month
  Peak diastolic flow velocity

CONTACTS AND LOCATIONS:
Overall Officials: Allan Klein, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No